CLINICAL TRIAL: NCT01279447
Title: Infrapatellar Nerve Block for Post-operative Analgesia for Knee Arthroscopy
Brief Title: Infrapatellar Nerve Block for Post-operative Knee Arthroscopy Pain Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Larry Hsu, Resident, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00026632
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-01

CONDITIONS: Internal Derangement of Knee
Keywords: infrapatellar nerve; saphenous nerve; knee arthroscopy; nerve block
MeSH Terms: interventions — Bupivacaine; Nerve Block; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Sham Comparator): A sham infrapatellar block performed under US guidance with normal saline
  Interventions: Drug: Normal Saline
- Infrapatellar nerve block (Experimental): An infrapatellar nerve block performed under US guidance with 0.25% bupivacaine
  Interventions: Drug: 0.25% Bupivacaine

INTERVENTIONS:
Drug: 0.25% Bupivacaine — 10cc, single dose, US guided injection
  Other Names: Nerve block
  Arms: Infrapatellar nerve block
Drug: Normal Saline — 10cc, single dose, US guided injection
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether infrapatellar branch of the saphenous nerve blocks are effective in decreasing analgesic use, promoting earlier mobility, and improving long term outcome scores after knee arthroscopy.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether infrapatellar branch of the saphenous nerve blocks are effective in decreasing analgesic use, promoting earlier mobility, and improving long term outcome scores after knee arthroscopy. Randomized, double-blinded, placebo controlled, study.

ELIGIBILITY:
Inclusion Criteria:

* planned knee arthroscopy with soft tissue intervention
* age 18+
* English speaking

Exclusion Criteria:

* contraindications to nerve block: eg neuropathy, type 1 diabetes, coagulopathy
* knee arthroscopy with planned bony intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Nuber, MD, Principal Investigator — Northwestern University; Antoun Nader, MD, Study Director — Northwestern University; Lawrence Hsu, MD, Study Director — Northwestern University; Mark Kendall, MD, Study Director — Northwestern University
Locations (1):
- Olson Surgical Pavilion, Chicago, Illinois, United States

REFERENCES:
- [Background] Akkaya T, Ersan O, Ozkan D, Sahiner Y, Akin M, Gumus H, Ates Y. Saphenous nerve block is an effective regional technique for post-menisectomy pain. Knee Surg Sports Traumatol Arthrosc. 2008 Sep;16(9):855-8. doi: 10.1007/s00167-008-0572-4. Epub 2008 Jun 24. PMID 18574578
- [Background] Lundblad M, Kapral S, Marhofer P, Lonnqvist PA. Ultrasound-guided infrapatellar nerve block in human volunteers: description of a novel technique. Br J Anaesth. 2006 Nov;97(5):710-4. doi: 10.1093/bja/ael241. Epub 2006 Sep 26. PMID 17005509
- [Background] Arthornthurasook A, Gaew-Im K. Study of the infrapatellar nerve. Am J Sports Med. 1988 Jan-Feb;16(1):57-9. doi: 10.1177/036354658801600110. PMID 3344881

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Infrapatellar Nerve Block
Started | 34 | 34
Completed | 31 | 33
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Population: Both groups statistically similar
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Infrapatellar Nerve Block | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (14.1) | 51.7 (12.1) | 50.6 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 18 | 15 | 33

OUTCOME MEASURES:

1. Primary Outcome: Post op Pain Score
Description: immediate postop pain score, Visual Analog Scale. Evaluates pain on scale from 0-10. 0=no pain. 10=maximum pain.
Time Frame: 0 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Infrapatellar Nerve Block
Number analyzed (Participants) | 34 | 34
units on a scale | 5.5 (2.6) | 3.9 (3.3)

ADVERSE EVENTS:
Arm/Group | Placebo | Infrapatellar Nerve Block
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34

LIMITATIONS AND CAVEATS:
outpatient nature and self reporting of outcome measures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes